CLINICAL TRIAL: NCT00809874
Title: Effects of Dietary Proteins on Postprandial Lipaemia and Incretin Responses in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: The Danish Obesity Research Centre (Other); Nordic Centre of Excellence (Other); Arla Foods (Industry)
Responsible Party: Kjeld Hermansen, Professor, Chief Physician, MD, Dr.Med.Sci, Department of Endocrinology And Metabolism, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CERN-PPL-JHJ
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Postprandial Lipaemia; Postprandial Incretins; Postprandial Inflammation
Keywords: Postprandial Period; Postprandial Lipaemia; Incretins; Subclinical Inflammation; Obesity; Atherosclerosis; Triglyceride; Lipoproteins
MeSH Terms: conditions — Obesity; Atherosclerosis | interventions — Caseins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Casein (Active Comparator)
  Interventions: Dietary Supplement: Casein
- Whey Isolate (Active Comparator)
  Interventions: Dietary Supplement: Whey Isolate
- Whey Hydrolysate (Active Comparator)
  Interventions: Dietary Supplement: Whey Hydrolysate
- Alphalact-Albumin (Active Comparator)
  Interventions: Dietary Supplement: Alphalact-Albumin

INTERVENTIONS:
Dietary Supplement: Casein
  Arms: Casein
Dietary Supplement: Whey Isolate
  Arms: Whey Isolate
Dietary Supplement: Whey Hydrolysate
  Arms: Whey Hydrolysate
Dietary Supplement: Alphalact-Albumin
  Arms: Alphalact-Albumin

SUMMARY:
The purpose of this study is to determine the effects of dietary protein on blood lipids and gut hormones after a fat-rich meal.

Hypothesis: Certain dietary proteins reduce the amount of fat circulating in the blood stream following a fat rich meal. The effect is dependant of both the quality and the quantity of protein ingested.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30 kg/m2 & <45 kg/m2

Exclusion Criteria:

* Diabetes
* lipid lowering drugs
* Liver-, Kidney- and/or Heart Disease
* Serious Hypertension (160/110)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Triglyceride | 0h- 1h- 2h- 4h- 6h- 7h- 8h postprandial

SECONDARY OUTCOMES:
Incretins | 0h -1h -2h -4h -6h -7h -8h Postprandial

CONTACTS AND LOCATIONS:
Overall Officials: K Hermansen, Professor, MD, Principal Investigator — Department of Endocrinology and Metabolism, Aarhus University Hospital
Locations (1):
- Department of Clinical Nutrion, Aarhus, Denmark